CLINICAL TRIAL: NCT04758676
Title: Bioelectric Impedance Analysis (BIA) Assessment of Polymyoneuropathy in Critically Ill Patients as a Part of Post-ICU Syndrome
Brief Title: BIA Assessment of Polymyoneuropathy in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Ostrava (Other)
Collaborators: University of Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KARIM-BIA-Ka21
Record Dates: First submitted 2021-01-14; First posted 2021-02-17 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Sepsis; Trauma; Respiratory Insufficiency; Surgery
Keywords: polymyoneuropathy; bioelectric impedance; post-intensive care syndrome; multiple organ dysfunction
MeSH Terms: conditions — Sepsis; Wounds and Injuries; Respiratory Insufficiency; postintensive care syndrome | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: There are two arms in the study - experimental group (diagnostics with the Multiscan 5000 device, nutritional recommendations, physiotherapy protocol), and control group (standard of care)
Masking Description: No masking is used in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional and physiotherapy protocol, BIA (Experimental): Study subjects randomized into this study arm will be indicated for nutritional and physiotherapy protocol, based upon the obtained results of the measurements, using bioimpedance analysis.
  Interventions: Other: Nutritional and physiotherapy protocol, BIA
- Standard of care (Active Comparator): Study subjects randomized into this study arm will be provided the current standard of care.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Nutritional and physiotherapy protocol, BIA — Study subjects will be treated using the nutritional and physiotherapy protocol, based upon the results of measurements, using bioimpedance analysis.
  Arms: Nutritional and physiotherapy protocol, BIA
Other: Standard of care — Study subjects will receive the current standard of care.
  Arms: Standard of care

SUMMARY:
The aim of the study is to monitor and evaluate changes in body composition, with a special emphasis on muscle mass, in the context of polyneuromyopathy of critically-ill patients at ICU, on artificial ventilation (duration of artificial ventilation at least 7 days), and subsequent comparison with the patient's condition in 12 weeks, as a part of Post-Intensive Care Syndrome (PICS) monitoring. The effect of the package (nutritional recommendations + physiotherapy protocol vs. standard of care) will be evaluated.

DETAILED DESCRIPTION:
Intensive medicine keeps pushing its borders, and enables survival of critical illnesses, including the substitution of organ functions in patients with multiple organ dysfunction (MODS). Despite the improvements in short-term outcomes, the long-term prognosis and quality of life (long-term outcomes) in patients, who survived a critical condition at ICU, remain unfavorable. The long-term consequences may persist for months or even years.

Post-intensive care syndrome (PICS) represents a significantly limiting impairment in three areas: physical (polyneuromyopathy of critically-ill patients), cognitive (delirium), and mental (development of depressions and PTSD - post-traumatic stress disorder). It is especially the rapid deterioration of muscles caused with the catabolic effect of the illness itself during accentuated proteolysis, very negatively affects the muscle strength, inability to discontinue artificial ventilation in the patient, increase of infections, and prolongation of the ICU stay. It often results in the inability to discharge the patient into home care. Polyneuromyopathy affects up to 40% of critically-ill patients; at the greatest risk are especially patients in a serious catabolic state, with activated systemic inflammatory response, with microvascular ischemia, on corticosteroids, immobilized, and on long-term artificial ventilation. The prevention is difficult, as well as monitoring of the lean body mass (LBM), especially in the muscle mass of critically ill patients, who are further affected with changes in hydration and fluid leak.

BIA - bioelectric impedance is a non-invasive technique, which is able, on the basis of impedance, to evaluate body composition (muscles, fat, total body fluid), determine hydration (ratio of extracellular and intracellular fluid, fluid retention); another prognostic marker is also the phase angle. It helps to evaluate markers of nutrition, basal energetic metabolism.

The BIS Multiscan 5000 device measures 50 frequencies, which are used to create a Cole Plot, using a mathematical model. It enables obtaining data from bed-ridden critically-ill patients, using tetrapolar bioelectric impedance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with respiratory insufficiency
* Expected period of artificial ventilation of 7 days
* Acute lung injury (ALI)
* Acute respiratory distress syndrome (ARDS)
* Acute exacerbation of chronic obstructive pulmonary disease (COPD)
* Signed informed consent (may be signed by witnesses, if the patient is unconscious)

Exclusion Criteria:

* Patients with unfavorable prognosis for 12-week follow-up
* APACHE Score >30
* Metastasizing malignity
* Patients after cardiopulmonary resuscitation (CPR) prior to admission
* Cerebral edema
* Cerebral trauma
* Intracranial hypertension
* Liver cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Body composition | 12 weeks
  Body composition will be studied using bioimpedance analysis - comparison of skeletal muscle mass, fats, body fluids

SECONDARY OUTCOMES:
Changes in the albumin level | 12 weeks
  Changes in the albumin level will be observed (in grams/Litre)
Changes in the prealbumin level | 12 weeks
  Changes in the prealbumin level will be observed (in milligrams/Litre)
Changes in the C-reactive protein (CRP) level | 12 weeks
  Changes in the C-reactive protein (CRP) level will be observed (in milligrams/Litre)
Changes in the presepsin level | 12 weeks
  Changes in the presepsin level will be observed (in picograms/millilitre)
Comparison of muscle functions | 12 weeks
  Comparison of muscle functions will be performed using dynamometry.

OTHER OUTCOMES:
Functional limitations - time up and go test (TUG) | 12 weeks
  Functional limitations will be assessed with TUG (time up and go test) (in seconds)
Functional limitations - spirometry - forced vital capacity (FCV) | 12 weeks
  Functional limitations will be assessed with spirometry - forced vital capacity (FCV) (volume)
Functional limitations - spirometry - forced expiratory velocity (FEV1) | 12 weeks
  Functional limitations will be assessed with spirometry - forced expiratory velocity in one second (FEV1) (velocity)
Cognitive state | 12 weeks
  Cognitive state of study subjects will be assessed with the presence of post-traumatic stress disorder (PTSD)

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Káňová, MD, Ph.D., Principal Investigator — University Hospital Ostrava
Locations (2):
- Czechia (2):
  - University of Ostrava, Department of Physiology and Patophysiology, Ostrava, Moravian-Silesian Region
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Derived] Kanova M, Petrekova K, Borzenko N, Ruskova K, Nytra I, Dzurnakova P, Burda M, Konvicka J. Bioelectrical Impedance in Monitoring Hyperhydration and Muscle Wasting in Critically Ill Corona Virus Disease (COVID-19) Patients: The Feasibility of Predicting Outcome. Physiol Res. 2025 Dec 31;74(Suppl 1):S93-S106. doi: 10.33549/physiolres.935748. PMID 41511101